CLINICAL TRIAL: NCT07397858
Title: Studies of Cognition and Behavior Using Sham Accelerated Transcranial Magnetic Stimulation
Brief Title: Cognition and Behavior With Sham Accelerated TMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Maitri Khanna, Co-Principal Investigator, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2375938
Record Dates: First submitted 2025-12-11; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
Keywords: TMS; Sham TMS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label sham (Other): All study participants will receive sham TMS (no active stimulation will be provided).
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Sham — All study participants will receive sham TMS (no active stimulation will be provided).

SUMMARY:
The goal of this clinical study is to understand how a person's expectations about treatment can influence their mood, motivation, and reactions to everyday rewards. The study includes young people ages 15-25 who will complete a sham (placebo) version of an accelerated transcranial magnetic stimulation (TMS) treatment. No active brain stimulation is given.

The main questions this study aims to answer are:

1. Do expectancy and treatment beliefs change during and after an accelerated sham TMS schedule?
2. Do these expectations influence mood, reward processing, or craving?
3. Does a more intensive schedule of sham sessions lead to different expectancy effects than a slower, once-daily schedule?

Participants will:

* Complete baseline clinical assessments and an MRI session
* Undergo five days of accelerated sham TMS (no active brain stimulation is delivered)
* Complete post-treatment MRI and follow-up assessments at 1 week and 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Able to provide informed consent (and assent if < 18 years)
* 15-25 years old

Exclusion Criteria:

* Unable to consent (due to medical condition, psychosis, substance use, etc)
* Acute suicidal crisis or with active medical illness that would interfere with participation
* Contraindications to receiving MRI as determined by screening questionnaires (Contraindications for MRI include metal in the body related to an injury or surgery, for example, surgical clips, metal fragments in the eyes, or piercings that cannot be removed. Subjects with braces or permanent retainers will not be scanned, because the effects on image signal are not well understood and may affect comparability between subjects and scan sites. Participants will be excluded for major neurological problems, such as seizure disorder, traumatic brain injury with loss of consciousness, or sensory problems that may impair task performance, such as blindness.)
* Participation in any clinical study with exposure to any investigational treatment or product within the previous 30 days, or plan on concurrent participation in other studies

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Accelerated sham TMS feasibility | From enrollment to end of study at 5 weeks
  Proportion of participants who complete the accelerated sham TMS protocol, defined as completion of all scheduled stimulation sessions. Feasibility will be assessed using session attendance logs and protocol completion records.
Change in treatment expectancy and beliefs | From enrollment to end of study at 5 weeks
  Change in treatment expectancy and beliefs score from baseline to end of study at 5 weeks, as measured by the Credibility/Expectancy Questionnaire (CEQ). Outcomes will be quantified as the difference in total CEQ score between time points. CEQ scores range from 1 to 9 for treatment credibility and expectancy, with higher scores indicating greater perceived credibility/ expectancy.
Change in reward sensitivity | From enrollment to end of study at 5 weeks
  Change in reward sensitivity will be assessed as the difference in scores from baseline to 5-week follow-up on validated self-report measures, including the Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ), the Snaith-Hamilton Pleasure Scale (SHAPS), and the Temporal Experience of Pleasure Scale (TEPS). SPSRQ scores range from 0-24 for each subscale, TEPS scores range from 18-108, and SHAPS scores range from 14-56, with higher scores indicating greater sensitivity to reward/punishment, pleasure capacity, and anhedonia, respectively.
Change in craving and engagement | From enrollment to end of study at 5 weeks
  Changes in cravings and engagement with reinforcing stimuli will be assessed as the difference in scores from baseline to 5-week follow-up on various self-report measures and tasks. Craving will be assessed using a behavioral craving task, with outcomes quantified as change in task-derived craving ratings or performance metrics from baseline to follow-up. Substance use will additionally be assessed as change in drug use frequency and quantity over the study period.

SECONDARY OUTCOMES:
Changes in depressive symptoms | From enrollment to end of study at 5 weeks
  Change in depressive symptoms will be measured as the difference in total score from baseline to 5-week follow-up on the Montgomery-Asberg Depression Rating Scale (MADRS). MADRS scores range from 0-60, with higher scores indicating greater depressive symptom severity.
Changes in mania symptoms | From enrollment to end of study at 5 weeks
  Change in mania symptoms will be measured as the difference in total score from baseline to 5-week follow-up on the Young Mania Rating Scale (YMRS). YMRS scores range from 0-60, with higher scores indicating greater manic symptom severity.
Changes in suicidality | From enrollment to end of study at 5 weeks
  Suicidality will be assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS), with changes evaluated based on trajectories and patterns of ideation and behavior responses from baseline to the 5-week follow-up. Higher response levels reflect greater suicidality symptom severity.
Change in quality of life and functioning | From enrollment to end of study at 5 weeks
  Change from baseline in quality of life and functional outcomes, assessed using the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF), a standardized self-report measure evaluating satisfaction and functioning across multiple life domains. Q-LES-Q-SF scores range from 14-70, with higher scores indicating greater quality of life and satisfaction.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and secondary outcome measures will be shared in accordance with the Institutional Review Board, including demographic variables, symptom rating scale scores, treatment assignment indicators, and visit-level timepoint data. Direct identifiers will not be shared.